CLINICAL TRIAL: NCT01777230
Title: The Value of Preoperative Sentinel Lymph Node Mapping by Pelvic MR Lymphangiography and SPECT-CT in Cervical Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Unable to get required research materials
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Ronald Zweemer, Gynaecological oncologist, UMC Utrecht
Other Study IDs: NL43062.041.13
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no biospecimens are to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Alle subjects included retain in one cohort.
  Interventions: Procedure: SPECT-CT sentinel node mapping; Procedure: Magnetic Resonance Lymphangiography sentinel node mapping; Procedure: Intra-operative sentinel node procedure

INTERVENTIONS:
Procedure: SPECT-CT sentinel node mapping — sentinel node localisation using the nuclear medicine technique SPECT-CT
  Other Names: Single Photon Emission Computed Tomography; Computed Tomography
Procedure: Magnetic Resonance Lymphangiography sentinel node mapping — Sentinel node localisation using Magnetic Resonance Lymphangiography
Procedure: Intra-operative sentinel node procedure — Open or (robot-assisted) laparoscopic sentinel node detection and resection.

SUMMARY:
Objective of the study: To study the concordance of sentinel node (SN) localization between preoperative Magnetic Resonance Lymphangiography and SPECT-CT SN mapping and the intra-operative SN procedure for low stage cervical cancer.

Background: The SN procedure for surgically treated cervical cancer is promising. Unfortunately, efficient and direct intra-operative SN localisation, without an extensive surgical exploration, remains a challenge even with combined use of patent blue dye en technetium-99m (99mTc). Preoperative imaging (= mapping) with 99mTc based SPECT-CT, which is increasingly adopted, has partly alleviated this problem. The investigators aim to investigate the feasibility of a new SN mapping modality, which visualises the (sentinel) lymph nodes using a Magnetic Resonance Imaging (MRI) technique (so called; Magnetic Resonance Lymphangiography), and compare it to SPECT-CT.

Design: Prospective, feasibility type diagnostic study. 40 subjects targeted. Via vaginal speculum exam, a specific MRI contrast-agent will be intracervically injected. Subsequently, on a wide bore 1.5T MRI system multiplanar imaging is performed, followed by a blinded review (experienced radiologist) for bilateral SN localization. Standard care with a preoperative SPECT-CT (after intracervical 99mTc administration). A blinded nuclear medicine specialist will localize the SN on the SPECT-CT images. Open or (robot-assisted) laparoscopy performed for localization of the blue stained and/or 99mTc-hot SN. Excision of the SN with freeze sectioning and histological review. Statistical analysis with intrapatient testing for concordance of MR Lympangiography and SPECT-CT based SN localization against the reference standard: the intra-operative sentinel node procedure.

DETAILED DESCRIPTION:
Background of the study: The sentinel procedure (SN) for surgically treated cervical cancer is promising. Unfortunately, efficient and direct intra-operative SN localisation, without an extensive retroperitoneal exploration, remains a challenge even with combined use of patent blue dye en 99mTc. The draining lymph nodes are positioned around the retroperitoneal pelvic vasculature, in close relation to the ureters and nerves innervating bladder, rectum and sexual functionality (inferior hypogastric plexus, genitofemoral nerve, etc), which makes exploration hazardous and time consuming. Furthermore, complete retroperitoneal exploration often necessitates dissection of lymph vessels (to find the SN) which would have been spared in a selective SN excision. The use of technetium-99m(99mTc) enables preoperative SN mapping with SPECT(-CT) to localise SN and partly alleviate this issue. Some clinics perform preoperative SPECT(-CT), despite its disadvantages of prolonged hospital admission, radiation exposure, limited spatial resolution (SPECT) and the limited soft tissue differentiation in the female pelvis (CT). The investigators postulate that Magnetic Resonance (MR) Lymphangiography is a better technique for preoperative SN mapping in cervical cancer. It allows for integration with regular work-up pelvic MRI and could make SPECT-CT unnecessary.

Objective of the study: To study the concordance of sentinel node localization between preoperative MR Lymphangiography and SPECT-CT SN mapping and the intra-operative sentinel node procedure (patent blue and 99mTc) for low stage cervical cancer.

Study design: Prospective, feasibility type diagnostic study with the experimental test (MR Lymphangiography) added to standard clinical care (SPECT-CT, intra-operative SN procedure).

Methods: 40 subjects targeted. Via a vaginal speculum exam 1ml of MR contrastmedium will be intracervically injected peripheral of the cervical tumor at 3, 6, 9 and 12 o'clock (suspine position). On a wide bore digital 1.5T MRI multiplanar T1w imaging is performed, followed by a blinded review (experienced radiologist) for bilateral SN localization with a standardized anatomical system. Standard procedure with a preoperative 220 MBq 99mTc SPECT-CT, a blinded nuclear medicine specialist will localize the SN. Standard peri-operative care; under general anesthesia 1ml injection of patent blue V in each of the four quadrants. Open or (robot-assisted) laparoscopy performed for visual localization of the blue SN's. Introduction of a gamma-probe and localization 'hot and blue' SN. For both methods anatomical locations of the SN are registered. Excision SN for freeze sectioning and histological review. Statistical analysis with intrapatient testing for concordance of SPECT-CT and MR Lympangiography based SN localization against the reference standard: the intra-operative sentinel node procedure (Patent blue and 99mTc).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary malignancy of the cervix uteri;
2. Primary therapy is surgery with minimally an intra-operative SN procedure and pelvic lymph node dissection;
3. ≥18 years of age and written inform consent provided.

Exclusion Criteria:

1. Contra-indications to MR lymphangiography, defined as:

   * All MRI incompatible electronic and/or ferromagnetic objects;
   * Presence of any object in the pelvic area prohibiting good image quality;
   * Severe claustrophobia;
   * Pregnancy or breastfeeding;
   * Unable to lie still and in complete supine position for 45 minutes;
   * Body weight >150kg;
   * History of an allergic reaction to any gadolinium based contrast agent;
   * Renal disease with a glomerular filtration rate (GFR) ≤ 30 mL/min/1.73m2;
2. History of an allergic reaction to patent blue V dye;
3. Any type of neo-adjuvant chemo and/or radiotherapy for cervical cancer;
4. Altered anatomy of pelvic lymph nodal drainage system (e.g. history of retroperitoneal pelvic surgery or trauma).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically proven cervical cancer which are a candidate for surgery, which includes an intra-operative SN procedure and pelvic lymph node dissection. Subjects are derived form a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Level of concordance in sentinel node (SN) localization between Magnetic Resonance Lymphangiography and SPECT-CT SN mapping with the intra-operative SN detection (based on blue dye and Tc-99m-nanocolloid). | within 1 week

SECONDARY OUTCOMES:
The absolute number of SN detected and uni/bilateral SN detection rates by MR lymphangiography, SPECT-CT, intra-operative SN procedure with patent blue only and combined patent blue / 99mTc. | within 1 week
The false negative rates in SN localization by MR lymphangiography, SPECT-CT, intra-operative SN procedure with patent blue only and combined patent blue / 99mTc. | within 1 week
Disagreement between the; concordance SN localization SPECT-CT and intra-operative SN procedure (blue + 99mTc) with the concordance MR lymphangiography and intra-operative blue dye only SN procedure (strategy without 99mTc). | within 1 week
  The difference in concordance (imaging to intra-operative results) between two strategies are compared.
  * The 1st strategy entails preoperative imaging with SPECT-CT and 'standard' intra-operative SN procedure (= with 99mTc use).
  * The 2nd strategy is with preoperative MR lymphangiography and an intra-operative 'blue dye only' SN procedure (= without 99mTc).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Zweemer, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands